CLINICAL TRIAL: NCT00656435
Title: Bevacizumab Pretreatment and Long Acting Gas Infusion on the Vitreous Clear-up After Diabetic Vitrectomy
Brief Title: Bevacizumab and Long Acting Gas in Diabetic Vitrectomy
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Chung-May Yang/Department of Opthalmology, National Taiwan University Hospital, Department of Opthalmology, National Taiwan University Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 200709051M
Record Dates: First submitted 2008-03-30; First posted 2008-04-11 (Estimated); Last update posted 2008-04-11 (Estimated); Status verified 2008-02

CONDITIONS: Proliferative Diabetic Retinopathy
Keywords: proliferative diabetic retinopathy; bevacizumab (Avastin); vitreous hemorrhage; long acting gas
MeSH Terms: conditions — Vitreous Hemorrhage | interventions — Bevacizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- A (Experimental): Patients will receive intravitreal injection of 1.25 mg of bevacizumab (0.05 ml) 7 to 9 days before vitrectomy
  Interventions: Drug: Bevacizumab
- B (No Intervention): Patients will not receive bevacizumab pretreatment

INTERVENTIONS:
Drug: Bevacizumab — Patients will receive intravitreal injection of 1.25 mg of bevacizumab (0.05 ml) 7 to 9 days before vitrectomy
  Other Names: Avastin
  Arms: A

SUMMARY:
Persistent or recurrent vitreous hemorrhage after vitrectomy for diabetic retinopathy complications is a common occurrence with an incidence of 12% to 63%. This complication may prolong vitreous clear-up and delay visual rehabilitation significantly, and sometimes requires additional procedures or surgery.

The causes of bleeding are diverse. Evidence suggests fibrovascular proliferation from the sclerotomy sites or from the vitreous base may be an important source of recurrent vitreous hemorrhage; other sources of bleeding include iatrogenic intraoperative injury of retinal vessels, and incomplete removal of fibrovascular tissues.

We have reported on the possible benefit of peripheral retinal cryotherapy and cryotherapy treatment of sclerotomy sites to prevent delayed-onset recurrent vitreous hemorrhage, and the possible benefit of intravitreal long-acting gas to reduce the occurrence of early postoperative recurrent vitreous hemorrhage, especially for cases with active fibrovascular proliferation. However, minor recurrent vitreous hemorrhage and prolonged reabsorption of lysed blood clots from surgical trauma remain important factors to cause media opacity long enough to prevent quick visual rehabilitation.

Intravitreal bevacizumab has been noted to induce rapid regression of retinal and iris neovascularization in proliferative diabetic retinopathy. Further, presurgical administration of intravitreal bevacizumab may reduce intraoperative bleeding during membrane dissection in PDR with traction retinal detachment. We hypothesize that presurgical treatment of intravitreal bevacizumab may reduce intraoperative bleeding and the amount of residual blood clots, while intraoperative infusion of long-acting gas may facilitate post-operative recovery of surgically injured retinal vessels. These combined effects would thus enhance early clear-up of vitreous opacity from clot lysis and recurrent retinal bleeding. To investigate this hypothesis, a clinical prospective study was undertaken to evaluate the effects of bevacizumab pretreatment combined with intravitreal infusion of long-acting gas on the clearance speed and the recurrence rate of early postoperative vitreous hemorrhage in vitrectomy for active diabetic fibrovascular proliferation.

DETAILED DESCRIPTION:
From December 2006 to August 2007, consecutive patients undergoing primary pars plana vitrectomy for active proliferative diabetic retinopathy were recruited for the prospective study. Included cases should have active fibrovascular proliferation with vitreo-retinal adhesions in 3 or more sites but not extending beyond equator in more than one quadrant. Active fibrovascular proliferation is defined as visible new vessels within the proliferative membranes with any degree of fresh vitreous or preretinal hemorrhage. Exclusion criteria are: 1. History of preoperative or postoperative anticoagulant therapy; 2. History of blood diseases associated with abnormal coagulation; 3. Severe proliferation with anticipation of silicone oil usage. Informed consent is obtained in every patient before surgery. The protocol was approved by the review board and research ethics committee of National Taiwan University Hospital.

All cases in the study group are prospectively enrolled (group 1). Consecutive patients fulfilling the enrollment criteria receive intravitreal bevacizumab (1.25mg in 0.05ml) injection 7 to 9 days before surgery and intravitreal 10% C3F8 infusion at the end of surgery. The surgical outcomes are compared with a non-concurrent control group that received gas infusion only (group2). The control group is matched by baseline characteristics and the severity of diabetic proliferation with the study group. The comparisons between the two groups are possible because all the relevant parameters have been carefully documented in the control group. A single surgeon (CMY) performed all of the operations.

Operative Technique For intravitreal bevacizumab injection, after topical anesthesia, patients were disinfected three times with povidone-iodine solution and draped. After eyelid speculum put in place, the eyes are further anesthetized with proparacaine -soaked cotton-tip applicators. Bevacizumab (1.25mg in 0.05ml) is drawn into a 1 ml syringe through a 27-gauged needle from a newly opened vial and injected through a 30-gauged needle into the vitreous cavity via temporal lower pars plana. Anterior chamber paracentesis is not performed.

Standard 3-port pars plana vitrectomy as described previously is done in every case. In short, vitreoretinal traction, fibrovascular tissues, and opacified vitreous as well as blood clots adherent to the peripheral vitreous skirt are removed as completely and safely as possible. Hemostasis is obtained by raising the infusion bottle, mechanical compression using a soft-tipped cannula, endodiathermy, or a combination of the above techniques. Blood clots formed during tissue dissection are removed carefully except on the bleeding sites where they were trimmed to small islands. Panretinal photocoagulation in non-laser treated eyes or supplementary laser in previously laser-treated eyes extending beyond the level of the equator is performed. Further peripheral retinal cryotherapy (10 to 12 spots in one row) is done. 10% C3F8 intravitreal infusion is done in each case before wound closure. Finally, cryotherapy of the sclerotomy sites (1 spot, each 6 seconds, for 3 sclerotomy sites) is performed.

After surgery, all patients are kept in a prone position overnight, and maintained a head-down position during waking hours. The patients are then allowed to lie on either side during sleep for 3 weeks thereafter. Ophthalmological examinations are performed in the first 4 days after surgery, then weekly for 4 weeks, biweekly for 1 month, and then monthly for at least 6 months.

The preoperative, intraoperative, and postoperative data are collected for each patient. These demographics and clinical findings included age, gender, study eye, types, duration and treatment regiment of diabetes mellitus, systemic diseases such as hypertension, renal insufficiency, intraoperative diagnosis, extent of vitreo-retinal adhesion, degree of intraoperative bleeding, duration of the surgery, and combined lens extraction. The extent of neovascularization, the severity of retinal traction, and the amount of fresh vitreous hemorrhage before and one week after bevacizumab injection were documented and, if possible, photographed. Data regarding the duration for vitreous clear-up; the time, duration, frequency and treatment of recurrent vitreous hemorrhage; and the duration of postoperative follow-up are also compiled. The extent of fibrovascular proliferation is graded as follows: grade 1, focal adhesions only; grade 2, broad adhesion ≥ one site(s) or vitreous-retinal adhesion at the disc, macula, and arcade; and grade3, vitreous-retinal attachment extending to the periphery. Intraoperative bleeding is classified into 3 grades : grade 1, minor bleeding that stopped either spontaneously or by transient bottle elevation; grade 2, moderate bleeding requiring endodiathermy or with formation of broad sheets of clots extending away from the bleeding site; grade 3, thick clot formation covering at least half of the posterior pole or interfering with the surgical plane.

Results of ophthalmological examinations, including best corrected visual acuity, intraocular pressure, lens status, and intravitreal gas amount, are recorded. We define vitreous clear-up time (VCUT) as the interval between the end of the surgery and the time when visualization of retinal vessels regained below the gas bubble. VCUT equal to or more than 3 weeks is considered prolonged. We define recurrent vitreous hemorrhage as recurrent hemorrhage that obscured the retinal vessels (grade 2 or above in the Diabetic Retinopathy Vitrectomy Study14) for more than one week after VCUT. Both early (≤ 4 weeks) and late (> 4weeks) recurrent vitreous hemorrhage are recorded. The severity of vitreous hemorrhage was classified according to the scale defined in the Diabetic Retinopathy Vitrectomy Study, and is reconfirmed by another ophthalmologist for every patient. The VCUT, the rate and treatment of recurrent vitreous hemorrhage, and the change of best-corrected visual acuity were compared between groups 1 and 2. Visual acuity is graded into three levels: low (≤1 meter counting fingers), moderate (>1 meter counting fingers, but < 20/200), and good (≥ 20/200).

Statistical Analysis To examine the differences among groups 1 and 2, discrete variables are performed statistical analysis with chi-squared test or Fisher's exact test. Continuous variables are presented as mean ± standard deviation and the Wilcoxon rank sum test was performed to make comparisons among groups 1 and 2. To further verify the effect of combined bevacizumab and gas treatment and to examine other possible factors affecting vitreous clear-up time, we would perform multivariate logistic regression analysis to determine the significance of the following factors: age, gender, duration of diabetes (< 10 years or ≥ 10 years), treatment regiment of diabetes, prior pan-retinal photocoagulation, hypertension, renal insufficiency, extent of fibrovascular proliferation, duration of surgery, and intravitreal bevacizumab. All of the statistical analyses are performed using STATA 8.2 software (StataCorp LP, College Station, Texas, USA). A P value < 0.05 was considered statistically significant.

ELIGIBILITY:
Inclusion Criteria:

1. anticoagulant therapy has not been used prior to surgery or during post-operative follow-up period.
2. no medical history of blood diseases associated with abnormal blood coagulation is present.
3. Having active fibrovascular proliferation with vitreo-retinal adhesions in 3 or more sites but not extending beyond the equator in more than one quadrant.
4. Severe retinopathy with anticipation of silicone oil usag
5. Age is between 20 to 85 years old.

Exclusion Criteria:

1. Not primary pars plana vitrectomy
2. post-operative follow-up duration less than three months
3. Pregnancy
4. HbA1c > 8.0

Ages: 20 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2006-12; Primary Completion 2007-08 (Actual); Study Completion 2008-02 (Actual)

PRIMARY OUTCOMES:
The severity of intraoperative bleeding and vitreous clear-up time. | Six months

SECONDARY OUTCOMES:
Percentage of prolonged vitreous clear-up (≥ 3 weeks) and recurrent hemorrhage rate. | Six months

CONTACTS AND LOCATIONS:
Overall Officials: Chung-May Yang, MD, Principal Investigator — National Taiwan University Hospital
Locations (1):
- Department of Ophthalmology, National Taiwan University Hospital, Taipei, Taiwan